CLINICAL TRIAL: NCT04800237
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy and Safety of VQW-765 in Patients With Performance Anxiety
Brief Title: Evaluating the Effects of VQW-765 vs. Placebo in Performance Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VQW-765-2201
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Performance Anxiety
Keywords: social phobia; social anxiety disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VQW-765 (Experimental)
  Interventions: Drug: VQW-765
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VQW-765 — oral capsule
  Arms: VQW-765
Drug: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of a single oral dose of VQW-765 compared to placebo in male and female participants with performance anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent.
* Sufficiently fluent in English to participate in the trial.
* Male and female patients aged 18-70 years (inclusive).

Exclusion Criteria:

* Lifetime history of bipolar disorder, schizophrenia, psychosis, seizures, delusional disorders or obsessive-compulsive disorder.
* Current or planned pregnancy or nursing during the trial period.
* A positive test for substances of abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | 1 Day

SECONDARY OUTCOMES:
Clinician Global Impression of Change (CGI-C) scale at visit 2 | 1 Day
Patient Global Impression of Change (PGI-C) scale at visit 2 | 1 Day
Assessment of safety and tolerability of a single dose of VQW-765, as measured by spontaneous reporting of adverse events (AEs) | 1 Day

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Vanda Investigational Site, Tempe, Arizona
  - Vanda Investigational Site, Beverly Hills, California
  - Vanda Investigational Site, Garden Grove, California
  - Vanda Investigational Site, San Jose, California
  - Vanda Investigational Site, Torrance, California
  - Vanda Investigational Site, Orlando, Florida
  - Vanda Investigational Site, Boston, Massachusetts
  - Vanda Investigational Site, North Dartmouth, Massachusetts
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Berlin, New Jersey
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, Staten Island, New York
  - Vanda Investigational Site, Raleigh, North Carolina
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No